CLINICAL TRIAL: NCT03709472
Title: Computer Assisted Family Intervention to Treat Self- Harm Disparities in Latinas and Sexual/Gender Minority Youth (CA CIFFTA)
Brief Title: Computer Assisted Family Intervention to Treat Self-Harm Disparities in Latinas and Sexual/Gender Minority Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Victoria Mitrani, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170791; U54MD002266 (NIH)
Record Dates: First submitted 2018-10-05; First posted 2018-10-17 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Self Harm; Depression; Emotion Dysregulation; Suicidal Ideation; Family Relations
MeSH Terms: conditions — Self-Injurious Behavior; Depression; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Randomization will be stratified by gender, type of self-harm, trauma exposure and LGBT status. The investigators will attempt to match overall contact hours (in the experimental condition some of these hours will be with technology). During the "continuing care" phase the CIFFTA families will interact with the therapist via the website for a period of 8 additional weeks. To match dosage time during aftercare, Treatment As Usual (TAU) will receive "check-in" telephone calls with the therapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer Assisted CIFFTA (Experimental): CA CIFFTA (Computer Assisted Culturally Informed and Flexible Family Based Treatment for Adolescents) consists of a hybrid intervention utilizing office-based CIFFTA and technology-delivered material. Over 16 weeks CIFFTA participants receive 45 minutes of face-to-face sessions plus approximately 45 minutes of web-based intervention per week. During the continuing care phase participants access website resources and receive targeted messages (e.g., handling family conflicts). CA CIFFTA will: 1) deliver psycho-educational modules (e.g., depression, emotion regulation), 2) collect diary-card information, and 3) provide additional resources. During videos parents and adolescents can report symptoms and information that is automatically transmitted to therapists and used in the next session
  Interventions: Behavioral: Computer Assisted CIFFTA
- Behavioral: Traditional face-to-face treatment-no technology (Active Comparator): Participants randomized to Treatment-As-Usual (TAU) work over a 16-week period with their community agency. They may receive individual or family treatment. The team coordinates with the TAU agencies to minimize the overlap of data collected. The team will refer out to service locations that are most convenient for the participant. A great deal of thought has gone into the selection of the Treatment as Usual condition. The investigators wanted to compare CA CIFFTA's ability to retain and bring about change in participants with what is typically done in the community. Although running an in-house comparison condition gives more control of the delivery of services and tracking of clients, it is difficult to know how that compared to the services that are typically provided in the community
  Interventions: Behavioral: Behavioral: Traditional face-to-face treatment-no technology

INTERVENTIONS:
Behavioral: Computer Assisted CIFFTA — This is a hybrid intervention that includes individual work with the adolescent (e.g., Motivational Interviewing, diary card identification of triggers), computer assisted psychoeducational work, and intensive family therapy interventions.
  Other Names: Behavioral: Family Therapy; Behavioral: Individual Therapy; Behavioral: Technology delivered psycho-educational modules
  Arms: Computer Assisted CIFFTA
Behavioral: Behavioral: Traditional face-to-face treatment-no technology — Community agencies provide mostly individual counseling but may add some family involvement in treatment planning.
  Other Names: Behavioral: Individual Therapy; Behavioral: Family Therapy
  Arms: Behavioral: Traditional face-to-face treatment-no technology

SUMMARY:
This study is designed to refine and test the efficacy of a computer assisted culturally informed and flexible/adaptive intervention for Latino adolescents for whom self-harm behaviors are a health disparity-specifically, Latinas and sexual/gender minority youth.

DETAILED DESCRIPTION:
This study enhances an original Computer Assisted Culturally Informed and Flexible Family-Based Treatment for Adolescents (CA CIFFTA) to directly address key targets related to self-harm behavior (e.g., depression, emotion dysregulation, LGBT, culture-related stressors, and trauma-related stressors); (b) refines the technological aspects of CA CIFFTA for web-based delivery; and (c) tests the preliminary efficacy of the new intervention and its delivery system in a randomized trial of 100 Hispanic adolescents and their parents. The investigators seek to reduce risk for repeated self-harm by showing treatment effects on depression, emotion regulation, substance use, and family functioning. Participants are randomly assigned to CA CIFFTA or Treatment-As-Usual and treatment covers a four month period.

ELIGIBILITY:
Inclusion Criteria. The adolescent must:

* be 11 to 18 years old;
* self-report an act of self-harm in the past 6 months,
* meet criteria for cut-off on two of the four underlying/maintaining factors (depression, emotion dysregulation, family conflict, substance use), and
* live with at least one parent-figure who agrees to participate in assessments and treatment Participants should be willing and able to participate fully in the protocol (e.g., to accept assignment to either condition, to provide sufficient locator information for follow-up, to allow their treatment sessions to be recorded for fidelity/process assessment and supervision).

Exclusion Criteria. Youth who:

* have a history of DSM V Developmental Disorders, Elective Mutism, Organic Mental Disorders, Schizophrenia, Delusional Disorder, Psychotic Disorder, and Bipolar Affective Disorder.
* are actively in crisis and reporting current ideation with a specific plan and with means to complete the plan.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 172 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Santisteban, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Institute for Individual and Family Counseling, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For each family, an adolescent and a caregiver were consented and participated in the study. 42 adolescents and their caregivers were randomized in each arm and received intervention. However, for the outcome measures section, only the adolescent's data was collected and reported for the study.
Pre-assignment Details: Four families declined to participate after enrollment (consent and intake assessment) and before randomization.
Period: Baseline
Arm/Group | Computer Assisted CIFFTA | Behavioral: Traditional Face-to-face Treatment-no Technology
Started | 84 | 84
Adolescent | 42 | 42
Caregiver | 42 | 42
Completed | 84 | 84
Not Completed | 0 | 0
Period: 4 Month Assessment (Post Treatment)
Arm/Group | Computer Assisted CIFFTA | Behavioral: Traditional Face-to-face Treatment-no Technology
Started | 84 | 84
Adolescent | 38 | 27
Caregiver | 38 | 27
Completed | 76 | 54
Not Completed | 8 | 30
Not completed — Lost to Follow-up | 8 | 30
Period: Assessment (12-month Post Baseline)
Arm/Group | Computer Assisted CIFFTA | Behavioral: Traditional Face-to-face Treatment-no Technology
Started (For each assessment time point, the 4-month post treatment assessment and the 12-month assessment, all participants were invited to complete the assessment even if they did not complete the previous time period. For this reason, the number of participants at the start of each arm is 84.) | 84 | 84
Adolescent | 36 | 19
Caregiver | 36 | 19
Completed | 72 | 38
Not Completed | 12 | 46
Not completed — Lost to Follow-up | 12 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computer Assisted CIFFTA | Behavioral: Traditional Face-to-face Treatment-no Technology | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 42 | 84
  Between 18 and 65 years | 42 | 42 | 84
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Adolescents and Caregivers reported separately for this analysis
  Participants
    Adolescent: number analyzed (Participants) | 42 | 42 | 84
    Adolescent: Female | 38 | 34 | 72
    Adolescent: Male | 4 | 6 | 10
    Adolescent: Intersex | 0 | 1 | 1
    Adolescent: Unknown | 0 | 1 | 1
    Caregiver: number analyzed (Participants) | 42 | 42 | 84
    Caregiver: Female | 39 | 37 | 76
    Caregiver: Male | 3 | 5 | 8
    Caregiver: Intersex | 0 | 0 | 0
    Caregiver: Unknown | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Adolescents and Caregivers reported separately for this analysis
  Participants
    Adolescent: number analyzed (Participants) | 42 | 42 | 84
    Adolescent: Hispanic or Latino | 36 | 37 | 73
    Adolescent: Not Hispanic or Latino | 3 | 2 | 5
    Adolescent: Unknown or Not Reported | 3 | 3 | 6
    Caregiver: number analyzed (Participants) | 42 | 42 | 84
    Caregiver: Hispanic or Latino | 38 | 40 | 78
    Caregiver: Not Hispanic or Latino | 4 | 2 | 6
    Caregiver: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Adolescents and Caregivers reported separately for this analysis
  Participants
    Adolescent: number analyzed (Participants) | 42 | 42 | 84
    Adolescent: American Indian or Alaska Native | 4 | 1 | 5
    Adolescent: Asian | 0 | 1 | 1
    Adolescent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Adolescent: Black or African American | 1 | 3 | 4
    Adolescent: White | 25 | 26 | 51
    Adolescent: More than one race | 0 | 0 | 0
    Adolescent: Unknown or Not Reported | 12 | 11 | 23
    Caregiver: number analyzed (Participants) | 42 | 42 | 84
    Caregiver: American Indian or Alaska Native | 0 | 0 | 0
    Caregiver: Asian | 0 | 0 | 0
    Caregiver: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregiver: Black or African American | 2 | 0 | 2
    Caregiver: White | 8 | 7 | 15
    Caregiver: More than one race | 0 | 0 | 0
    Caregiver: Unknown or Not Reported | 32 | 35 | 67

OUTCOME MEASURES:

1. Primary Outcome: Columbia Suicide Severity Rating Scale (CSSRS) Suicide Ideation
Description: The Columbia yields information on suicide ideation and Ideation with Intent. Youth were categorized as having or not having ideation and having or not having intent to suicide (yes/no). Endorsing any of these items as "yes" is a worse outcome. The number listed below is the number of participants that said "yes" to experiencing suicidal ideation in the last month.
Time Frame: Baseline, 4 months post baseline, 12 months post baseline
Population: Only data from adolescents was collected. Missing data is because they did not provide sufficient item responses to calculate a score. Participants can respond with "don't know" or "refuse". This interferes with scoring.
Measure: Count of Participants; unit: Participants
Arm/Group | Computer Assisted CIFFTA | Behavioral: Traditional Face-to-face Treatment-no Technology
Number analyzed (Participants) | 38 | 27
Participants
  Baseline: number analyzed (Participants) | 36 | 26
  Baseline | 20 | 13
  4-month assessment (post-treatment): number analyzed (Participants) | 36 | 24
  4-month assessment (post-treatment) | 16 | 8
  12-month assessment (12 months post baseline): number analyzed (Participants) | 31 | 18
  12-month assessment (12 months post baseline) | 6 | 4

2. Secondary Outcome: Number of Participants Who Reported Self-harm Behavior
Description: The Deliberate Self-harm Inventory Youth Version (DSHI-Y) documents self-harm behavior. The data collected focused on the number of participants who reported "yes" to having engaged in self-harm in the past 30 days.
Time Frame: Baseline, 4 months post baseline, 12 months post baseline
Population: Only data from adolescents was collected. Missing data is because they did not provide sufficient item responses to calculate a score. Participants can respond with "don't know" or "refuse" and this interferes with scoring.
Measure: Count of Participants; unit: Participants
Arm/Group | Computer Assisted CIFFTA | Behavioral: Traditional Face-to-face Treatment-no Technology
Number analyzed (Participants) | 38 | 27
Participants
  Baseline: number analyzed (Participants) | 38 | 26
  Baseline | 25 | 18
  4- month assessment (post treatment assessment): number analyzed (Participants) | 36 | 24
  4- month assessment (post treatment assessment) | 14 | 11
  12 months assessment (12 months post baseline): number analyzed (Participants) | 33 | 17
  12 months assessment (12 months post baseline) | 4 | 4

3. Secondary Outcome: Emotional Dysregulation Measured by Emotion Regulation Scale -Short Form (DERS)
Description: Difficulties with Emotion Regulation Scale -Short form (DERS), is designed to assess emotional dysregulation using a 5-point Likert Scale. The total score is calculated from the sum of all items, with higher scores indicating greater problems with emotion regulation. Total summed scores can range from 18 - 90 but investigators report that average item score (1-5) rather than the sum so that is more easily interpretable in the 5 point Likert Scale.
Time Frame: Baseline, 4 months post baseline, 12 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Computer Assisted CIFFTA | Behavioral: Traditional Face-to-face Treatment-no Technology
Number analyzed (Participants) | 38 | 27
score on a scale
  Baseline: number analyzed (Participants) | 38 | 26
  Baseline | 3.1 (.75) | 3.2 (.78)
  4-month assessment (post-treatment) | 2.8 (.59) | 2.9 (.78)
  12-month assessment post baseline: number analyzed (Participants) | 36 | 19
  12-month assessment post baseline | 2.6 (.76) | 2.8 (.71)

4. Secondary Outcome: The Patient Health Questionnaire
Description: The PHQ-9 incorporates the DSM-IV depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool. Depression Severity: 0 - none, 1-4 minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Time Frame: Baseline, 4 months post baseline, 12 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Computer Assisted CIFFTA | Behavioral: Traditional Face-to-face Treatment-no Technology
Number analyzed (Participants) | 38 | 27
score on a scale
  Baseline | 13.9 (6.3) | 14.9 (7.0)
  4-month assessment (post treatment): number analyzed (Participants) | 36 | 24
  4-month assessment (post treatment) | 10.8 (5.8) | 11.6 (7.7)
  12-month assessment (12 months post baseline): number analyzed (Participants) | 34 | 19
  12-month assessment (12 months post baseline) | 8.9 (6.7) | 10.9 (7.7)

5. Secondary Outcome: Family Connectedness
Description: The Family Connectedness (FC) scale includes seven items assessing communication and the relationship between parents and youth. A composite score was obtained. Two items measured communication and five items measured connectedness. The five Items were scored on a 1-10 scale and summed to a total connectedness score. Minimum score = 5 and Maximum score = 50. Higher scores mean better connections.
Time Frame: Baseline, 4 months post baseline, 12 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Computer Assisted CIFFTA | Behavioral: Traditional Face-to-face Treatment-no Technology
Number analyzed (Participants) | 32 | 23
score on a scale
  Baseline | 32.1 (9.3) | 28.4 (10.5)
  4-month assessment (post treatment) | 33.4 (8.8) | 31.4 (10.6)
  12-month assessment (12 months post baseline): number analyzed (Participants) | 32 | 19
  12-month assessment (12 months post baseline) | 32.1 (11.3) | 30.2 (9.5)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Only adolescent data was collected for adverse events.
Arm/Group | Computer Assisted CIFFTA | Behavioral: Traditional Face-to-face Treatment-no Technology
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

LIMITATIONS AND CAVEATS:
The COVID disruptions reduced our overall sample size. A limitation is that we did not collect dosage data on treatment received by TAU participants. Finally, with only two timepoints and a small sample, it was impossible to analyze mediation. The best we could do was to explore plausible mediators (Emotion Regulation and Family Connectedness).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT03709472/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT03709472/SAP_001.pdf
  • Informed Consent Form (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT03709472/ICF_002.pdf